CLINICAL TRIAL: NCT03552510
Title: Impact of Oro-Pharyngeal Administration of Mother's Milk Prior to Gavage Feeding on GIT Motility in Preterm Infants
Brief Title: Oropharyngeal Administration of Mother's Milk in Preterm Infants and Gastrointestinal Motility
Acronym: OPAMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nehad Nasef, Professor of Pediatrics, Mansoura University Children Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS.15.06.01
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Preterm Infant; Feeding Disorder Neonatal; Gastrointestinal Motility Disorder
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Oropharyngeal Administration of mother's milk (OPAMM)
Who Masked: Outcomes Assessor
Masking Description: Laboratory assessment of GIT hormonal level will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial OPAMM (Active Comparator): At the start of the study, infants will receive mother's milk (to the maximum of 0.2 ml) to the oro-pharyngeal pouch, tongue and cheeks every 3 hours (5 minutes before time of feeding), and the remaining amount will be given by regular gavage feeding for 24 hours.
  Then, infants will receive regular gavage feeding only for the next 24 hours.
  Interventions: Procedure: Oro-pharyngeal Administration of Mother's Milk
- Initial Gavage (Active Comparator): At the start of the study, infants will receive regular gavage feeding only for 24 hours.
  Then, infants will receive mother's milk (to the maximum of 0.2 ml ) by dropper to the oro-pharyngeal pouch, tongue and cheeks every 3 hours (5 minutes before time of feeding), and the remaining amount will be given by regular gavage feeding for the next 24 hours.
  Interventions: Procedure: Oro-pharyngeal Administration of Mother's Milk

INTERVENTIONS:
Procedure: Oro-pharyngeal Administration of Mother's Milk — Infants will receive mother's milk (to the maximum of 0.2 ml ) by dropper to the oro-pharyngeal pouch, tongue and cheeks every 3 hours (5 minutes before time of feeding)

SUMMARY:
Mother's milk does not come in contact with the oropharyngeal pouch of preterm infants during gavage feeding. We hypothesized that stimulation of the oropharyngeal pouch using small amount of the mother's milk 5 minutes before initiation of regular gavage feeding will increase the level of GIT hormones.

DETAILED DESCRIPTION:
Feeding preterm infants continues to challenge health care providers because of difficulty to provide adequate volume of milk that maintains optimum nutrition without increasing the risk of feeding intolerance. Preterm, VLBW, infants are at increased risk of feeding intolerance as they have shorter GIT with lower digestive, absorptive, and motility capabilities than those of full-term infants. Intolerance to enteral feeding has been associated with abdominal distention, initiation of inflammatory cascade, edema of the bowel, and subsequent development of necrotizing enterocolitis.

Oral feeding is the best physiologic method for enteral nutrition of preterm infants. However, because of immaturity of suckling reflex and poor coordination between suckling and swallowing, gavage feeding (oro-gastric or naso-gastric tube feeding) has been used an alternative method of enteral nutrition in preterm infants.

During breastfeeding, mother's milk comes in contact with mouth and oro-pharyngeal pouch which, theoretically, stimulates both oro-pharyngeal receptors that improves the motility, secretory, and absorptive ability of the GIT. Furthermore, anti-inflammatory and pro-inflammatory cytokines, which are present abundantly in mother's colostrum and milk, may exert an immuno-protective effect when they come in contact with oro-pharyngeal as well as GIT mucosa.

Preterm, VLBW, infant in the NICU receives enteral feedings by a naso-gastric or oro-gastric gavage tube. Thus, mother's milk does not typically come into contact with oro-pharyngeal pouch which delays the maturation of oral suckling and swallowing skills in preterm infants.

Oral stimulation has been shown to improve oral feeding performance, attain early oral feeding, improve weight gain and shorten the length of hospital stay. Investigators aimed to study the effect of Oro-pharyngeal administration of mother's milk before regular gavage feeding on gastrointestinal movement in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants delivered at less than 32 weeks gestation and less than 1500 grams birth weight will be included in the study

Exclusion Criteria:

1. Preterm infants > 32 weeks gestation unable to be fed on own mother's colostrum or milk.
2. Preterm infants with major congenital anomalies or chromosomal abnormalities.
3. Preterm infants delivered to mothers with confirmed chorioamnionitis.
4. Preterm infants with confirmed early onset sepsis.

Ages: 1 Day to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Motilin hormone | 24 hours
  Plasma Motilin hormone level
Gastrin hormone | 24 hours
  Plasma Gastrin hormone level
Secretin hormone | 24 hours
  Plasma Secretin hormone level
Cholecystokinin | 24 hours
  Plasma Cholecystokinin hormone level

SECONDARY OUTCOMES:
Feeding residual | 24 hours
  Percentage of feeding residual after each fed
Holding feeds | 24 hours
  Frequency of withholding feeds for suspected feeding intolerance

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, El Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided